CLINICAL TRIAL: NCT03199703
Title: Randomized Trial of Conventional Versus Radiofrequency Needle Transseptal Puncture for Cryoballoon Ablation
Brief Title: Conventional Versus RF Needle Transseptal Puncture for Cryoballoon Ablation
Acronym: CRYO-LATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jason Andrade (Other)
Collaborators: Baylis Medical Company (Industry)
Responsible Party: Sponsor-Investigator, Jason Andrade, MD FRCPC FHRS, University of British Columbia
Organization: University of British Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6-May-16
Record Dates: First submitted 2017-06-09; First posted 2017-06-27 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Atrial Fibrillation
Keywords: PVI Ablation; Cryoballoon
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: 150 patients will be randomized in a 1:1, single-blinded fashion to 1 of 2 transseptal groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baylis transseptal system group (Active Comparator): Patients randomized to the Baylis transseptal system group (Bayliss Group) will undergo transseptal puncture with a large, preformed curve 71-cm-C1 or 98-cm-C1 18-gauge NRG needle (Baylis Medical) through a TorFlex sheath (Baylis Medical), with the sheath curve selected at the discretion of the operating physician.
  Interventions: Device: Baylis transseptal system group
- Conventional transseptal group (Active Comparator): Patients randomized to the conventional transseptal group (Standard Group) will undergo transseptal puncture with either a large, preformed curve 71- or 98-cm 18-gauge BRK needle (BRK, BRK-1, BRK-2 needle, St. Jude Medical) through any non-Baylis sheath (for example Schwartz SL, Biosense-Webster Preface) selected at the discretion of the operating physician.
  Interventions: Device: Standard conventional transseptal group

INTERVENTIONS:
Device: Baylis transseptal system group
  Arms: Baylis transseptal system group
Device: Standard conventional transseptal group
  Arms: Conventional transseptal group

SUMMARY:
This will be a prospective single-blinded, randomized, controlled trial comparing the effectiveness and safety of transseptal puncture using the Baylis transseptal system to transseptal left atrial access with standard transseptal equipment (usual care) in patients undergoing catheter ablation procedures for atrial fibrillation with the cryoballoon system.

The targeted population will consist of patients with symptomatic paroxysmal atrial fibrillation undergoing pulmonary vein isolation with the cryoballoon system.

DETAILED DESCRIPTION:
Study Objective - The objective of the prospective, randomized study is to evaluate the effectiveness and safety of the Baylis transseptal system (RF needle, TorFlex sheath, and specialised ProTrack guidewire) compared with a conventional transseptal (conventional sheath, Brockenbrough needle, and standard guidewire) for transseptal LA access during cryoballoon ablation procedures.

Trial design - This will be a prospective single-blinded, randomized, controlled trial comparing the effectiveness and safety of transseptal puncture using the Baylis transseptal system to transseptal left atrial access with standard transseptal equipment (usual care) in patients undergoing catheter ablation procedures for atrial fibrillation with the cryoballoon system.

Study Population - The targeted population will consist of patients with symptomatic paroxysmal atrial fibrillation undergoing pulmonary vein isolation with the cryoballoon system.

ELIGIBILITY:
Inclusion Criteria:

* Non-permanent AF documented on a 12 lead ECG, Trans Telephonic Monitoring (TTM) or Holter monitor within the last 24 months
* Age of 18 years or older on the date of consent
* Candidate for ablation based on AF that is symptomatic
* Informed Consent

Exclusion Criteria:

* Previous left atrial (LA) ablation or LA surgery
* AF due to reversible cause (e.g. hyperthyroidism, cardiothoracic surgery)
* Active Intracardiac Thrombus
* Pre-existing pulmonary vein stenosis or PV stent
* Pre-existing hemidiaphragmatic paralysis
* Contraindication to anticoagulation or radiocontrast materials
* Left atrial anteroposterior diameter greater than 5.5 cm by transthoracic echocardiography
* Cardiac valve prosthesis
* Clinically significant (moderately-severe, or severe) mitral valve regurgitation or stenosis
* Myocardial infarction, PCI / PTCA, or coronary artery stenting during the 3-month period preceding the consent date
* Cardiac surgery during the three-month interval preceding the consent date
* Significant congenital heart defect (including atrial septal defects or PV abnormalities but not including PFO)
* NYHA class III or IV congestive heart failure
* Left ventricular ejection fraction (LVEF) less than 35%
* Hypertrophic cardiomyopathy (septal or posterior wall thickness >1.5 cm)
* Significant Chronic Kidney Disease (CKD - eGFR <30 µMol/L)
* Uncontrolled hyperthyroidism
* Cerebral ischemic event (strokes or TIAs) during the six-month interval preceding the consent date
* Pregnancy
* Life expectancy less than one (1) year
* Currently participating or anticipated to participate in any other clinical trial of a drug, device or biologic that has the potential to interfere with the results of this study
* Unwilling or unable to comply fully with study procedures and follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Total time required for left atrial access | Intraprocedural assessment (within 24 hours)
  defined as time from the first pull-down of the needle/sheath/dilator apparatus in the superior vena cava to first entrance of the cryoballoon into the left atrium.

SECONDARY OUTCOMES:
Transeptal Access | Intraprocedural assessment (within 24 hours)
  Success/failure of the assigned transseptal apparatus to achieve transeptal puncture (proportion of patients necessitating the use of the alternate study apparatus - e.g. cross-over from the NRG RF needle to the to conventional BRK needle)
Plastic Shavings | Intraprocedural assessment of visible plastic shavings (within 24 hours)
  Proportion of cases whereby the presence (or absence) of visible plastic dilator shavings from needle introduction are seen
The proportion of patients sustaining a procedural complication plausibly related to transseptal puncture | Acute peri-procedural complications will be defined as occurring within 30 days of ablation
  Events include pericardial effusion, pericardial tamponade, cardiac perforation, air embolism, aortic root puncture
Transseptal time - septal engagement to sheath advancement | Intraprocedural assessment (measured in seconds)
  Time from inter-atrial septum engagement with the transseptal needle to FlexCath sheath advancement into the LA
Transseptal time - left atrial access to sheath positioning | Intraprocedural assessment (measured in seconds)
  Time from needle advancement through the septum to sheath advancement into the LA

CONTACTS AND LOCATIONS:
Locations (6):
- Canada (6):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, University of British Columbia, Vancouver, British Columbia
  - Queen Elizabeth II, Halifax, Nova Scotia
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Université Laval, Québec, Quebec
  - University of Saskatchewan, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Andrade JG, Macle L, Bennett MT, Hawkins NM, Essebag V, Champagne J, Roux JF, Makanjee B, Tang A, Skanes A, Khaykin Y, Morillo C, Jolly U, Lockwood E, Amit G, Angaran P, Sapp J, Wardell S, Wells GA, Verma A, Deyell MW. Randomized trial of conventional versus radiofrequency needle transseptal puncture for cryoballoon ablation: the CRYO-LATS trial. J Interv Card Electrophysiol. 2022 Nov;65(2):481-489. doi: 10.1007/s10840-022-01277-y. Epub 2022 Jun 24. PMID 35739438